CLINICAL TRIAL: NCT02649478
Title: A Randomized, Parallel-Group, Placebo-Controlled, Clinical Endpoint Bioequivalence Study of Generic Fluticasone Propionate 100 µg and Salmeterol Xinafoate 50 µg Inhalation Powder Compared With Advair Diskus® 100/50 in Subjects With Asthma
Brief Title: Clinical Endpoint Bioequivalence Study for Fluticasone Propionate and Salmeterol Xinafoate
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Roxane Laboratories (Industry)
Collaborators: Vectura Limited (Industry)
Responsible Party: Sponsor
Organization: West-Ward Pharmaceutical (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FLSA-P100/50-PVCL-1
Record Dates: First submitted 2016-01-05; First posted 2016-01-07 (Estimated); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Fluticasone-Salmeterol Drug Combination

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Fluticasone / Salmeterol (Experimental): fluticasone propionate (100 mcg) and salmeterol xinafoate (50 mcg) administered via the Vectura lever operated multidose inhaler ("LOMI") inhaler device twice a day by inhalation throughout the study
  Interventions: Drug: Fluticasone / Salmeterol
- Advair Diskus 100/50 (Active Comparator): Advair Diskus (fluticasone propionate and salmeterol xinafoate) twice a day by inhalation throughout the study
  Interventions: Drug: Advair Diskus 100/50
- placebo inhaler (Placebo Comparator): placebo inhaled powder twice a day by inhalation throughout the study
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fluticasone / Salmeterol — Fluticasone propionate (100 mcg) and salmeterol xinafoate (50 mcg) administered via the Vectura LOMI inhaler device
  Arms: Fluticasone / Salmeterol
Drug: Placebo
  Arms: placebo inhaler
Drug: Advair Diskus 100/50 — Advair (Fixed dose combination of Fluticasone propionate and salmeterol xinafoate administered via the Diskus inhaler device)
  Arms: Advair Diskus 100/50

SUMMARY:
A Randomized, Parallel-Group, Placebo-Controlled, Clinical Endpoint Bioequivalence Study of Generic Fluticasone Propionate 100 µg and Salmeterol Xinafoate 50 µg Inhalation Powder Compared with Advair Diskus® 100/50 in Subjects with Asthma

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the clinical bioequivalence of generic fluticasone propionate 100 µg and salmeterol xinafoate 50 µg inhalation powder (test) to Advair Diskus ("Advair") 100/50 (reference) for the treatment of asthma.

The secondary objectives of the study are:

* To demonstrate statistical superiority of generic fluticasone propionate 100 µg and salmeterol xinafoate 50 µg inhalation powder to placebo.
* To demonstrate statistical superiority of Advair 100/50 to placebo.
* To investigate the safety and tolerability of fluticasone propionate 100 µg and salmeterol xinafoate 50 µg inhalation powder compared with Advair 100/50 in the target population.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects must be 12 years of age or older. Females must be of non-childbearing potential or if of childbearing potential, must commit to consistent use of a form of birth control which is medically effective.
2. Be able to provide written informed consent or, in the case of adolescents, informed assent in addition to an informed consent form signed by the adolescent's parent(s) or legal guardian(s).
3. Be current non-smokers and also may not have used tobacco products (e.g., cigarettes, cigars, pipe tobacco) within the year prior to Visit 1, and have 10 years or less (10 pack-years for cigarettes) of historical use.
4. Have persistent asthma, as defined by the National Asthma Education and Prevention Program, for at least 12 weeks before Visit 1.
5. The forced expiratory volume at one second ("FEV1") range required for enrollment is dependent on whether the subject is an adult or adolescent and whether he or she is currently treated with inhaled corticosteroids ("ICS") at Visit 1
6. Demonstrate 15% or greater reversibility of FEV1 between 10 and 30 minutes following 360 µg of albuterol inhalation. NOTE: If the subject does not meet criterion 6 at Visit 1 (Day -14), this criterion must be met at Visit 2 (Day -1).
7. Be able to discontinue controller asthma medication (including leukotriene modifiers ("LTM"), ICS and long acting β-agonists (LABAs)) during the Run-in Period and Treatment Period.
8. Be able to replace current short-acting β-agonists (SABAs) with the study-supplied albuterol (or equivalent) rescue medication inhaler for use as needed for the duration of the study (subjects should be able to withhold all inhaled SABAs for a least 6 hours before lung function assessments during study visits).
9. Be appropriately using 1 of the following asthma-treatment regimens and meet the associated criteria:

   * Low- to medium-dose ICS for at least 4 weeks before Visit 1, with or without an adjunctive asthma therapy (i.e., LABA, LTM, or theophylline). Both the ICS dose and overall daily asthma regimen must have been stable for the 4 weeks before Visit 1; or
   * Leukotriene modifier (such as montelukast, zafirlukast, or pranlukast) or theophylline as monotherapy at a stable dose for at least 4 weeks before Visit 1;or
   * Daily (or near daily) rescue medication (e.g., albuterol/ salbutamol or other inhaled SABA used to treat acute asthma) in the 4 weeks before Visit 1.
10. Must not have been treated (for any reason) with oral or parenteral corticosteroids for at least 1 month before Visit 1 and must not have used oral SABAs for at least 12 hours before Visit 1 and for the remainder of the study. Routine use of oral/parenteral corticosteroids and oral SABAs is not allowed after Visit 1.
11. Subjects may continue using short-acting forms of theophylline (withheld at least 12 hours before a site visit), twice daily controlled release forms of theophylline (withheld at least 24 hours before a site visit), and once daily controlled-release forms of theophylline (withheld at least 36 hours before a site visit).
12. Be able to answer questions regarding asthma status and be able to document) device usage and asthma status on a twice daily basis.

    NOTE: Placebo inhaler use (i.e., compliance) must be at least 75% of the planned doses taken as assessed at Visit 2, for the subject to be considered eligible to continue in the study.
13. Demonstrate proper use of metered dose inhaler ("MDI") and dry-powder inhaler devices.

Exclusion Criteria:

1. Have an Asthma Control Questionnaire (ACQ) score of 3.0 or greater at Visit 1.
2. Are unable to discontinue ICS, LABA, or LTM.
3. Have a history of life-threatening asthma, defined as an asthma episode (at any time in the past) associated with any of the following: respiratory arrest or intubation, hypercapnia, hypoxic seizures, or syncopal episode.
4. Have exercise-induced asthma as the only asthma-related diagnosis that does not require daily asthma control medicine.
5. Have evidence or history of clinically significant disease or abnormality including congestive heart failure, uncontrolled hypertension, uncontrolled coronary artery disease, myocardial infarction, or cardiac dysrhythmia. In addition, historical or current evidence of significant hematologic, hepatic, neurologic, psychiatric, renal, or other diseases that in the opinion of the investigator, would put the subject at risk through study participation, or would affect the study analyses if the disease exacerbated during the study.
6. Have current clinical evidence of pneumonia, pneumothorax, atelectasis, pulmonary fibrotic disease, allergic bronchopulmonary aspergillosis, cystic fibrosis, bronchopulmonary dysplasia, chronic obstructive pulmonary disease, or other respiratory abnormalities other than asthma.
7. Have obstructive sleep apnea severe enough to require biphasic or continuous positive-airway pressure therapy, or likely to interfere with the assessment of asthma symptoms, in the investigator's judgment.
8. Using medication with the potential to affect the course of asthma or interact with sympathomimetic amines (e.g., β blockers [including eye drops], oral decongestants, benzodiazepines, digitalis, phenothiazines, polycyclic antidepressants, monoamine oxidase inhibitors).
9. Had a viral or bacterial, upper or lower respiratory tract infection or sinus or middle ear infection within 4 weeks before Visit 1 or have an infection during the Run-in Period.
10. Participated in an interventional study or used any investigational drug for any disease within 30 days (or 4 half lives, if this is longer than 30 days) before Visit 1 before Visit 1.
11. Used an anti-immunoglobulin E (e.g., omalizumab) or any other monoclonal antibody for any reason within 6 months before Visit 1.
12. Are hypersensitive to any β2-agonist sympathomimetic drug, or any intranasal, inhaled, or systemic corticosteroid therapy or any component of these combination medications including severe milk protein hypersensitivity.
13. Are exhibiting any factors (e.g., infirmity, disability, or geographic location, inability to follow instructions or study compliance requirements) that the investigator believes would likely limit the subject's compliance with the study protocol or scheduled site visits. This includes recent history of substance abuse or uncontrolled psychiatric or neurological behavior that would render the subject incapable of reliably following study requirements, in the judgment of the investigator.
14. Have an affiliation with the participating site; in other words, subject may not be an immediate family member of any study site staff and may not be employed directly or indirectly by the study site.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1430 (Actual)
Dates: Start 2014-08; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Baseline-adjusted area under the serial FEV1-time curve from time 0 to 12 hours on the first day of the Treatment Period | 0-12 hours after dosing on Day 1
Baseline-adjusted, pre-dose FEV1 on the last day of the Treatment Period | 30 Days

SECONDARY OUTCOMES:
Adverse Events | From Visit 1 (Day -28) until 30 days after the last dose of study drug

CONTACTS AND LOCATIONS:
Locations (100):
- United States (100):
  - Roxane Laboratories Research Site #30, Glendale, Arizona
  - Roxane Laboratories Research Site #46, Phoenix, Arizona
  - Roxane Laboratories Research Site #1, Surprise, Arizona
  - Roxane Laboratories Research Site #13, Tempe, Arizona
  - Roxane Laboratories Research Site #84, Bakersfield, California
  - Roxane Laboratories Research Site #72, Costa Mesa, California
  - Roxane Laboratories Research Site #67, Encinitas, California
  - Roxane Laboratories Research Site #4, Fountain Valley, California
  - Roxane Laboratories Research Site #64, Fullerton, California
  - Roxane Laboratories Research Site #3, Huntington Beach, California
  - Roxane Laboratories Research Site #70, Huntington Beach, California
  - Roxane Laboratories Research Site #92, Huntington Beach, California
  - Roxane Laboratories Research Site #38, Irvine, California
  - Roxane Laboratories Research Site #91, Lincoln, California
  - Roxane Laboratories Research Site #59, Los Angeles, California
  - Roxane Laboratories Research Site #16, Los Angeles, California
  - Roxane Laboratories Research Site #90, Los Angeles, California
  - Roxane Laboratories Research Site #6, Mission Viejo, California
  - Roxane Laboratories Research Site #78, Rolling Hills Estates, California
  - Roxane Laboratories Research Site #98, Sacramento, California
  - Roxane Laboratories Research Site #53, San Diego, California
  - Roxane Laboratories Research Site #93, San Diego, California
  - Roxane Laboratories Research Site #28, San Jose, California
  - Roxane Laboratories Research Site #60, Santa Monica, California
  - Roxane Laboratories Research Site #33, Centennial, Colorado
  - Roxane Laboratories Research Site #43, Denver, Colorado
  - Roxane Laboratories Research Site #63, Denver, Colorado
  - Roxane Laboratories Research Site #21, Wheat Ridge, Colorado
  - Roxane Laboratories Research Site #50, Hialeah, Florida
  - Roxane Laboratories Research Site #11, Hialeah, Florida
  - Roxane Laboratories Research Site #66, Homestead, Florida
  - Roxane Laboratories Research Site #83, Jupiter, Florida
  - Roxane Laboratories Research Site #8, Miami, Florida
  - Roxane Laboratories Research Site #23, Miami, Florida
  - Roxane Laboratories Research Site #86, Miami, Florida
  - Roxane Laboratories Research Site #89, Miami, Florida
  - Roxane Laboratories Research Site #20, Miami, Florida
  - Roxane Laboratories Research Site #68, Miami, Florida
  - Roxane Laboratories Research Site #80, Miami, Florida
  - Roxane Laboratories Research Site #54, Miami, Florida
  - Roxane Laboratories Research Site #12, Miami, Florida
  - Roxane Laboratories Research Site #74, North Miami Beach, Florida
  - Roxane Laboratories Research Site #35, Orlando, Florida
  - Roxane Laboratories Research Site #17, Orlando, Florida
  - Roxane Laboratories Research Site #94, Port Orange, Florida
  - Roxane Laboratories Research Site #34, Lilburn, Georgia
  - Roxane Laboratories Research Site #51, Rincon, Georgia
  - Roxane Laboratories Research Site #79, Normal, Illinois
  - Roxane Laboratories Research Site #47, River Forest, Illinois
  - Roxane Laboratories Research Site #100, Brownsburg, Indiana
  - Roxane Laboratories Research Site #62, Baltimore, Maryland
  - Roxane Laboratories Research Site #52, Baltimore, Maryland
  - Roxane Laboratories Research Site #71, Bethesda, Maryland
  - Roxane Laboratories Research Site #96, Silver Spring, Maryland
  - Roxane Laboratories Research Site #81, Fall River, Massachusetts
  - Roxane Laboratories Research Site #56, North Dartmouth, Massachusetts
  - Roxane Laboratories Research Site #55, Ann Arbor, Michigan
  - Roxane Laboratories Research Site #97, Chelsea, Michigan
  - Roxane Laboratories Research Site #5, Plymouth, Minnesota
  - Roxane Laboratories Research Site #85, St Louis, Missouri
  - Roxane Laboratories Research Site #32, Bellevue, Nebraska
  - Roxane Laboratories Research Site #25, Bellevue, Nebraska
  - Roxane Laboratories Research Site #36, Omaha, Nebraska
  - Roxane Laboratories Research Site #57, Las Vegas, Nevada
  - Roxane Laboratories Research Site #10, Atco, New Jersey
  - Roxane Laboratories Research Site #65, Skillman, New Jersey
  - Roxane Laboratories Research Site #7, New York, New York
  - Roxane Laboratories Research Site #2, New York, New York
  - Roxane Laboratories Research Site #41, Clemmons, North Carolina
  - Roxane Laboratories Research Site #45, Raleigh, North Carolina
  - Roxane Laboratories Research Site #31, Cincinnati, Ohio
  - Roxane Laboratories Research Site #95, Columbus, Ohio
  - Roxane Laboratories Research Site #24, Hilliard, Ohio
  - Roxane Laboratories Research Site #61, Middleburg Heights, Ohio
  - Roxane Laboratories Research Site #73, Toledo, Ohio
  - Roxane Laboratories Research Site #14, Edmond, Oklahoma
  - Roxane Laboratories Research Site #15, Oklahoma City, Oklahoma
  - Roxane Laboratories Research Site #37, Eugene, Oregon
  - Roxane Laboratories Research Site #40, Medford, Oregon
  - Roxane Laboratories Research Site #58, Portland, Oregon
  - Roxane Laboratories Research Site #26, Warwick, Rhode Island
  - Roxane Laboratories Research Site #99, Warwick, Rhode Island
  - Roxane Laboratories Research Site #69, Greenville, South Carolina
  - Roxane Laboratories Research Site #22, Spartanburg, South Carolina
  - Roxane Laboratories Research Site #19, Smyrna, Tennessee
  - Roxane Laboratories Research Site #27, Boerne, Texas
  - Roxane Laboratories Research Site #75, Dallas, Texas
  - Roxane Laboratories Research Site #49, El Paso, Texas
  - Roxane Laboratories Research Site #44, Houston, Texas
  - Roxane Laboratories Research Site #77, Lewisville, Texas
  - Roxane Laboratories Research Site #87, Plano, Texas
  - Roxane Laboratories Research Site #29, San Antonio, Texas
  - Roxane Laboratories Research Site #48, San Antonio, Texas
  - Roxane Laboratories Research Site #42, West Jordan, Utah
  - Roxane Laboratories Research Site #39, South Burlington, Vermont
  - Roxane Laboratories Research Site #9, Henrico, Virginia
  - Roxane Laboratories Research Site #88, Richmond, Virginia
  - Roxane Laboratories Research Site #18, Richmond, Virginia
  - Roxane Laboratories Research Site #76, Tacoma, Washington
  - Roxane Laboratories Research Site #82, Greenfield, Wisconsin